CLINICAL TRIAL: NCT00771875
Title: B-Cell Targeted Therapy for Acute Renal Allograft Rejection With an Antibody Mediated Component: A Prospective, Randomized, Open-Label Study
Brief Title: Randomized Trial for Mixed Acute Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, E. Steve Woodle, MD, FACS, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X05273
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Graft Rejection
MeSH Terms: interventions — thymoglobulin; Rituximab; Bortezomib; Acetaminophen; Histamine Antagonists; Diphenhydramine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rabbit Antithymocyte Globulin (RATG) (Active Comparator): Rabbit Antithymocyte Globulin (RATG) All patients will receive RATG (Thymoglobulin) dosed based on CD3 count. Patients will be redosed when the cluster of differentiation 3 (CD3) count is ≥ 25. Depending on rejection severity, Thymoglobulin will be given for a maximum of 7-14 days. CD3 levels will be monitored daily. 1.5mg/kg/day over 6 hrs with 1st dose (D1) and over 4 hours for each dose thereafter. (day 1 then when CD3 levels > 25 cells/mm3); Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care. Methylprednisolone 250 mg with 1st dose of Thymoglobulin. Methylprednisolone 125 mg on treatment day 2 subsequent corticosteroids per institution standard of care; following treatment, corticosteroid therapy will resume at the pre-rejection dose.
  Interventions: Drug: Rabbit Antithymocyte Globulin (RATG); Drug: Rituximab; Drug: Bortezomib; Drug: Acetaminophen; Drug: Antihistamine; Drug: Methylprednisolone
- RATG/Rituximab (Experimental): Rabbit Antithymocyte Globulin (RATG) + Rituximab Subjects will be given 1.5mg/kg/day of RATG over 6 hrs with 1st dose (D1) and over 4 hours for each dose thereafter. (day 1 then when CD3 levels > 25 cells/mm3); Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care. Rituximab dose of 375 mg/ m2 on day 2. Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care. Methylprednisolone 250 mg with 1st dose of Thymoglobulin. Methylprednisolone 125 mg on treatment day 2 subsequent corticosteroids per institution standard of care; following treatment, corticosteroid therapy will resume at the pre-rejection dose.
  Interventions: Drug: Rituximab; Drug: Acetaminophen; Drug: Antihistamine; Drug: Methylprednisolone
- RATG/Bortezomib (Experimental): Rabbit Antithymocyte Globulin (RATG) + Bortezomib -Subjects will be given 1.5mg/kg/day of RATG over 6 hrs with 1st dose (D1) and over 4 hours for each dose thereafter. (day 1 then when CD3 levels > 25 cells/mm3). Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care. Bortezomib will be given at a dose of 1.3 mg/m2 via IV push over 3-5 seconds on days 2, 5, 9, and 12. Methylprednisolone will be administered prior to each bortezomib dose. On days 2 and 5, administer methylprednisolone 100 mg intravenous push (IVP). On days 9 and 12, administer methylprednisolone 50 mg intravenous push (IVP). If thymoglobulin is administered the same day as bortezomib, the order of administration is- methylprednisolone, then bortezomib, then thymoglobulin.
  Interventions: Drug: Bortezomib; Drug: Acetaminophen; Drug: Antihistamine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Rabbit Antithymocyte Globulin (RATG) — All patients will receive Thymoglobulin dosed based on CD3 count. Patients will be redosed when the CD3 count is ≥ 25. Depending on rejection severity, Thymoglobulin will be given for a maximum of 7-14 days. CD3 levels will be monitored daily.
  Other Names: thymoglobulin
  Arms: Rabbit Antithymocyte Globulin (RATG)
Drug: Rituximab — Rituximab dose of 375 mg/ m2 on day 2. Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care.
  Other Names: rituxan
  Arms: RATG/Rituximab; Rabbit Antithymocyte Globulin (RATG)
Drug: Bortezomib — Patient will receive 1.3 mg/m2 via IV push over 3-5 seconds on days 2, 5, 9, and 12. Consolidation course of bortezomib will be dosed at 1.3 mg/m2 IVP X 4 doses administered on days 1, 4, 7 and 10.
  Other Names: Velcade
  Arms: RATG/Bortezomib; Rabbit Antithymocyte Globulin (RATG)
Drug: Acetaminophen — Patients will be premedicated with acetaminophen prior to dosing per institution standard of care.
  Other Names: Tylenol
Drug: Antihistamine — Patients will be premedicated with an antihistamine prior to dosing per institution standard of care.
  Other Names: diphenhydramine
Drug: Methylprednisolone — Methylprednisolone 250 mg with 1st dose of Thymoglobulin. Methylprednisolone 125 mg on treatment day 2 subsequent corticosteroids per institution standard of care; following treatment, corticosteroid therapy will resume at the pre-rejection dose.
  Other Names: Medrol

SUMMARY:
This study is being conducted to determine how safe and effective using an immune cell (b cell) depleting therapy and/or Thymoglobulin is in patients with a kidney transplant who are experiencing certain types of rejection.

DETAILED DESCRIPTION:
The purpose of the study is to determine safety and efficacy of treatment if mixed (cellular and antibody) mediated acute rejection with addition of B-cell depleting therapy to Thymoglobulin in kidney and simultaneous kidney pancreas allograft recipients.

ELIGIBILITY:
Inclusion Criteria

Each subject must meet all of the following inclusion criteria to be enrolled in the study:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use two acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Subject is between 18 and 65 years of age, inclusive.
* Subject has a transplant dysfunction indicated by an increase in creatinine of 0.3 mg/dL or 15% (lipase >3 X ULN for kidney/pancreas recipients) over baseline necessitating an allograft biopsy to assess for allograft rejection.
* Presence of light microscopic histologic changes consistent with acute cellular rejection of a Banff 97 (2005 update) grade IA or greater and at least one of the following:
* Donor-specific antibody (DSA) positive via Luminex
* Presence of C4d in the peritubular capillaries or glomeruli
* Subject must have no known contraindications to treatment with bortezomib, boron or mannitol, thymoglobulin, or rituximab.
* Recipients of kidney or simultaneous kidney pancreas organ transplant.

Exclusion Criteria

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study.

* Subject has a platelet count < 100,000/mm3 within 7 days before enrollment.
* Subject has an absolute neutrophil count of < 1,000/mm3 within 7 days before enrollment.
* Subject has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Subject has received other investigational drugs with 14 days before enrollment
* Serious medical (other than renal disease) or psychiatric illness likely to interfere with participation in this clinical study.
* Subjects that have previously received an organ transplant other than kidney or simultaneous kidney pancreas.
* Subjects who are recipients of A-B-O incompatible transplants, all cytotoxicity (CDC) crossmatch positive transplants
* Recipients of a simultaneous kidney pancreas transplant that only have pancreas rejection.
* Subjects unable to tolerate a dose of mycophenolate mofetil 1-3g/day (or equivalent mycophenolic acid dose).
* Subjects who are anti-HIV-positive, or HBsAg-positive. Anti-Hepatitis C Virus (HCV) positive patients are excluded, except patients with negative pathologic complete remission-result.
* Recipients of a kidney from a donor who tests positive for HIV, HBsAg or anti-HCV
* History of malignancy within the past 5 years that is not considered to be cured, with the exception of localized basal cell carcinoma of the skin (excised ≥ 2 years prior to randomization)
* Subjects with current or recent severe systemic infections within the 2 weeks prior to randomization.
* Receipt of a live vaccine within 4 weeks prior to study entry
* Evidence of severe liver disease with abnormal liver profile (aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin > 3 times upper limit of normal (ULN)) at screening.
* Pregnant or nursing (lactating) women.
* EBV sero-mismatch (EBV + donor organ transplanted to EBV - recipient)
* CMV sero-mismatch (CMV + donor organ transplanted to CMV - recipient)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Rabbit Antithymocyte Globulin (RATG): RATG
  Rabbit Antithymocyte Globulin (RATG): All patients will receive Thymoglobulin dosed based on cluster of differentiation 3 (CD3) count. Patients will be redosed when the CD3 count is ≥ 25. Depending on rejection severity, Thymoglobulin will be given for a maximum of 7-14 days. CD3 levels will be monitored daily.
  Rituximab: Rituximab dose of 375 mg/ m2 on day 2. Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care.
  Bortezomib: Patient will receive 1.3 mg/m2 via intravenous push (IVP) over 3-5 seconds on days 2, 5, 9, and 12. Consolidation course of bortezomib will be dosed at 1.3 mg/m2 IVP X 4 doses administered on days 1, 4, 7 and 10.
- RATG/Rituximab: Rabbit Antithymocyte Globulin (RATG) + Rituximab
  Rituximab: Rituximab dose of 375 mg/ m2 on day 2. Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care.
- RATG/Bortezomib: Rabbit Antithymocyte Globulin (RATG) + Bortezomib
  Bortezomib: Patient will receive 1.3 mg/m2 via IV push over 3-5 seconds on days 2, 5, 9, and 12. Consolidation course of bortezomib will be dosed at 1.3 mg/m2 IVP X 4 doses administered on days 1, 4, 7 and 10.
Period: Overall Study
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Started | 10 | 10 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rabbit Antithymocyte Globulin (RATG): RATG
  Rabbit Antithymocyte Globulin (RATG): All patients will receive Thymoglobulin dosed based on CD3 count. Patients will be redosed when the CD3 count is ≥ 25. Depending on rejection severity, Thymoglobulin will be given for a maximum of 7-14 days. CD3 levels will be monitored daily.
  Rituximab: Rituximab dose of 375 mg/ m2 on day 2. Patients will be premedicated with an antihistamine and acetaminophen prior to dosing per institution standard of care.
  Bortezomib: Patient will receive 1.3 mg/m2 via IV push over 3-5 seconds on days 2, 5, 9, and 12. Consolidation course of bortezomib will be dosed at 1.3 mg/m2 IVP X 4 doses administered on days 1, 4, 7 and 10.
- Total: Total of all reporting groups
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib | Total
Number analyzed (Participants) | 10 | 9 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (12.6) | 34.2 (6.6) | 38.5 (12.3) | 35.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 10
  Male | 8 | 5 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 10 | 29
Type of Transplant [Number; unit: participants]
  Deceased Donor Kidney Transplant | 2 | 1 | 3 | 6
  Deceased Donor Simultaneous Pancreas/Kidney | 1 | 1 | 2 | 4
  Living Donor | 7 | 7 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Group With Any of the Following: Rejection Reversal or Recurrent Rejection
Description: Rejection Reversal is a return of serum creatinine to within 115% of the baseline value, or histologic reversal occurring within 14 days of initiation of treatment.
  Recurrent Rejection is histologic evidence of rejection noted on a biopsy specimen obtained up to 3 months after documented rejection reversal.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
participants
  Rejection Recurrence | 0 | 0 | 0
  Rejection Reversal | 2 | 1 | 1

2. Secondary Outcome: Number of Patients With Allografts With C4d Focal Positive Pretreatment Biopsy
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
participants | 2 | 2 | 4

3. Secondary Outcome: Renal Allograft Survival
Time Frame: 1 year after rejection treatment
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
participants | 7 | 7 | 10

4. Secondary Outcome: Mean Serum Creatinine
Description: Renal allograft function as determined by change (∆) in Calculated creatinine clearance by Cockcroft-Gault at 7, 14, 28, 60, and 90 days and 1 year post therapy initiation
Time Frame: 7, 14, 28, 60, 90 days and 1 year post therapy initiation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
mg/dL
  7 days | 3.04 (1.67) | 2.32 (0.89) | 2.31 (0.78)
  14 days | 3.25 (1.76) | 2.35 (0.95) | 2.20 (0.69)
  28 days | 2.9 (1.23) | 2.35 (0.90) | 2.18 (0.47)
  60 days | 2.62 (1.23) | 2.32 (0.87) | 2.38 (0.62)
  90 days | 2.48 (1.18) | 2.12 (1.01) | 2.13 (0.54)
  1 year | 2.19 (0.84) | 2.07 (1.10) | 2.87 (1.37)

5. Secondary Outcome: Incidence of Death
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
participants | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Allografts With C4d Diffuse Positive Pretreatment Biopsy
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
participants | 3 | 3 | 5

7. Secondary Outcome: Incidence of Post Transplant Lymphoproliferative Disorder (PTLD)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Number analyzed (Participants) | 10 | 9 | 10
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rabbit Antithymocyte Globulin (RATG) | RATG/Rituximab | RATG/Bortezomib
Serious Adverse Events (participants affected / at risk) | 7/10 | 5/9 | 7/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabbit Antithymocyte Globulin (RATG) (N=10) | RATG/Rituximab (N=9) | RATG/Bortezomib (N=10)
Death due to hypoglycemic attack and respiratory distress (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pain and Tenderness at Pheresis Line (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 4 (4) | 5 (5)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Surgical Complication (Surgical and medical procedures) | 4 (4) | 1 (1) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Renal Dysfunction (Renal and urinary disorders) | 7 (19) | 5 (10) | 7 (20)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Serum Sickness (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Thombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage of Lower GI (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabbit Antithymocyte Globulin (RATG) (N=10) | RATG/Rituximab (N=9) | RATG/Bortezomib (N=10)
Grade 4 Thrombocytopenia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Grade 1 Nausea/Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2) | 5 (5)
Grade 2 Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2)
Grade 1 Diarrhea (Gastrointestinal disorders) | 6 (6) | 3 (3) | 3 (3)
Worsened Peripheral Neuropathy (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Grade 2 Anemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 3 (3)
Grade 3 Anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (5) | 2 (2)
Grade 4 Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus (CMV) infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BK Virus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tingling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Level 1 Peripheral Neuropathy (Renal and urinary disorders) | 5 (5) | 3 (4) | 4 (4)
Level 2 Peripheral Neuropathy (Renal and urinary disorders) | 0 (0) | 3 (3) | 4 (4)
Level 3 Peripheral Neuropathy (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Grade 2 Peripheral Neuropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Level 4 Peripheral Neuropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Level 5 Peripheral Neuropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes